CLINICAL TRIAL: NCT00350571
Title: Adaptive Brief Interventions for Drop-out Re-engagement
Brief Title: Brief Interventions for Drop-out Re-engagement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 101010101; 5P50DA009241-120012; 5P50DA009241 (NIH)
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Substance Abuse
Keywords: behavior therapy; counseling; drug abuse therapy; outpatient care; therapy compliance; clinical trial phase I; coping; outcomes research; satisfaction; social psychology; patient oriented research
MeSH Terms: conditions — Substance-Related Disorders; Patient Compliance; Personal Satisfaction | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care follow up (Active Comparator): Standard care counselor follow up care phone calls or letters.
  Interventions: Behavioral: standard care follow up
- Drop out reengagement motivational intervention (Experimental): Single session office based or phone based motivational counseling session designed to promote participant re-engagement in standard treatment.
  Interventions: Behavioral: brief (behavioral therapy); Behavioral: Drop out re-engagement motivational intervention

INTERVENTIONS:
Behavioral: brief (behavioral therapy) — up t 3 sessions of phone or office based counseling sessions to promote re-engagement in treatment.
  Arms: Drop out reengagement motivational intervention
Behavioral: Drop out re-engagement motivational intervention — Up to 3 phone or office based counseling sessions to promote reengagement in treatment
  Arms: Drop out reengagement motivational intervention
Behavioral: standard care follow up — routine counselor phone calls and letters
  Arms: Standard care follow up

SUMMARY:
We will evaluate a series of interventions intended to help individuals who drop out of substance abuse treatment re-engage in order to improve treatment outcome.

DETAILED DESCRIPTION:
We propose a 5-year Stage I behavioral therapy development study to: 1) prospectively evaluate risk factors for premature drop-out from outpatient treatment; 2) develop and test a manual of single session phone-and office-based interventions to re-engage these individual in treatment.

ELIGIBILITY:
Inclusion Criteria:

* admission to outpatient treatment

Exclusion Criteria:

* need for hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
retention into outpatient treatment | 4, 8, 12, 24 weeks

SECONDARY OUTCOMES:
substance abuse | 4, 8,12,and 24 weeks
psychiatric symptoms | 4, 8, 12, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ball, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - APT Foundation, New Haven, Connecticut
  - Connecticut Mental Health Center, New Haven, Connecticut